CLINICAL TRIAL: NCT03602482
Title: Standing Cognition and Co-morbidities of POTS Evaluation
Acronym: SCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Dysautonomia International (Other)
Responsible Party: Principal Investigator, Amanda Miller, Postdoctoral Fellow, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Study00009606
Record Dates: First submitted 2018-07-09; First posted 2018-07-26 (Actual); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Postural Tachycardia Syndrome; Ehlers-Danlos Syndrome
Keywords: postural tachycardia syndrome; cognition
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Ehlers-Danlos Syndrome | interventions — Standing Position; Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standing (Experimental): Participants will complete cognitive testing while standing.
  Interventions: Behavioral: Standing
- Supine (Active Comparator): Participants will complete cognitive testing while supine.
  Interventions: Behavioral: Supine

INTERVENTIONS:
Behavioral: Standing — Participants will stand and complete cognitive tests.
  Arms: Standing
Behavioral: Supine — Participants will complete cognitive tests while supine.
  Arms: Supine

SUMMARY:
The purpose of this study is to evaluate cognition in patients with postural tachycardia syndrome (POTS) while lying down and standing and to assess the prevalence of hypermobile Ehlers-Danlos Syndrome in POTS.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with POTS, or healthy control
* Age between 13-60 years
* Participants may be any race, ethnicity, sex, or gender
* Able and willing to provide informed consent

Exclusion Criteria:

* Inability to give, or withdrawal of, informed consent
* Age ≤ 13 or ≥ 61 years
* Prisoners
* Unable to stand

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 139 (Actual)
Dates: Start 2018-06-23 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda J Miller, Ph.D., Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 participants with POTS were recruited at the 2018 Dysautonomia International Conference in June 2018 in Nashville, TN.
  39 Healthy participants were enrolled at Penn State Hershey Medical Center from August 2018- December 2019,
Pre-assignment Details: Participants with odd study IDs completed cognitive testing while supine first. Participants with even study IDs completed cognitive testing standing first.
Groups:
- POTS- Supine First, Then Standing: Volunteers previously diagnosed with postural tachycardia syndrome, able to stand unassisted, age 13-60 years. Odd numbered participants assigned to complete cognitive tests in the supine posture first then in the standing posture.
- POTS- Standing First, Then Supine: Volunteers previously diagnosed with postural tachycardia syndrome, able to stand unassisted, age 13-60 years. Even numbered participants assigned to complete cognitive tests in the standing posture first, then supine.
- Controls- Supine First, Then Standing: Healthy volunteers with no chronic or systemic illness, age 13-60 years. Odd numbered participants assigned to complete cognitive tests in the supine posture first then in the standing posture.
- Controls- Standing First, Then Supine: Healthy volunteers with no chronic or systemic illness, age 13-60 years. Even numbered participants assigned to complete cognitive tests in the standing posture first, then supine.
Period: Overall Study
Arm/Group | POTS- Supine First, Then Standing | POTS- Standing First, Then Supine | Controls- Supine First, Then Standing | Controls- Standing First, Then Supine
Started | 50 | 50 | 20 | 19
Completed | 44 | 43 | 20 | 19
Not Completed | 6 | 7 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 7 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- POTS: Participants previously diagnosed with postural orthostatic tachycardia syndrome who were able to stand unassisted were enrolled
- Control: Healthy volunteers that were free of chronic illness were enrolled
- Total: Total of all reporting groups
Arm/Group | POTS | Control | Total
Number analyzed (Participants) | 100 | 39 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 2 | 17
  Between 18 and 65 years | 85 | 37 | 122
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [19 to 37] | 24 [23 to 29] | 25 [21 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 36 | 128
  Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 96 | 0 | 96
  Unknown or Not Reported | 0 | 39 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 96 | 35 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 100 | 39 | 139
education level [Mean (Standard Deviation); unit: years] | 15 (3) | 16 (2) | 15 (3)

OUTCOME MEASURES:

1. Primary Outcome: Executive Function (Stroop Word-color Test)
Description: Testing scores are normalized using T-scores for predicted values based on age and education for each participant. Scores range from 0 to 100. Higher numbers indicate better cognition. Testing will be performed while participants are supine and standing.
Time Frame: 1 hour
Population: 13 participants dropped out (by their choice) prior to study visit. Mean and standard deviation scores for each arm are reported.
Measure: Mean (Standard Deviation); unit: Testing Scores
Groups:
- POTS- Supine, Standing: Participants previously diagnosed with postural orthostatic tachycardia syndrome who were able to stand unassisted. Odd numbered participants were assigned to cognitive testing in the supine posture first, then in the standing posture.
- POTS- Standing, Supine: Participants previously diagnosed with postural orthostatic tachycardia syndrome who were able to stand unassisted. Even numbered participants were assigned to cognitive testing in the standing posture first, then in the supine posture.
- Control- Supine, Standing: Healthy volunteers that were free of chronic illness. Odd numbered participants were assigned to cognitive testing in the supine posture first, then in the standing posture.
- Control- Standing, Supine: Healthy volunteers, free of chronic illness. Even numbered participants were assigned to cognitive testing in the standing posture first, then in the supine posture.
Arm/Group | POTS- Supine, Standing | POTS- Standing, Supine | Control- Supine, Standing | Control- Standing, Supine
Number analyzed (Participants) | 44 | 43 | 20 | 19
Testing Scores
  Standing Stroop Scores | 48 (13) | 49 (10) | 50 (6) | 58 (9)
  Supine Stroop Scores | 45 (10) | 54 (12) | 55 (10) | 56 (10)

2. Secondary Outcome: Attention Score Using Cogstate Identification Task
Description: Scores are measured as speed to complete task with lower numbers indicating faster reaction time. Testing will be performed while participants are supine and standing.
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: reaction time (milliseconds)
Arm/Group | POTS- Supine, Standing | POTS- Standing, Supine | Control- Supine, Standing | Control- Standing, Supine
Number analyzed (Participants) | 44 | 43 | 20 | 19
reaction time (milliseconds)
  ID test speed standing | 2.78 (0.11) | 2.78 (0.12) | 2.70 (0.05) | 2.68 (0.06)
  ID test speed supine | 2.74 (0.09) | 2.64 (0.40) | 2.71 (0.06) | 2.70 (0.06)

3. Secondary Outcome: Number of Participants With Hypermobile Ehlers-Danlos Syndrome (hEDS)
Description: hEDS was evaluated using the Diagnostic Criteria for hEDS checklist. The number of participants who fulfill the diagnostic criteria on the checklist are reported.
Time Frame: 1 hour
Population: The number of participants who had hEDS are reported. This assessment was performed without respect to position (standing/supine) and only in POTS participants. Nine POTS participants did not complete this portion of the study. Healthy controls were not included in this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- POTS: POTS participants completed a screening for hypermobile EDS
Arm/Group | POTS
Number analyzed (Participants) | 91
Participants | 28

4. Secondary Outcome: Heart Rate Standing Minus Heart Rate Supine
Description: Heart rate (HR) will be measured using an arm blood pressure cuff while participants are in supine and standing postures. The difference in heart rate (HR standing - HR supine) was calculated for each participant.
Time Frame: 1 hour
Population: The change in heart rate (HR standing - HR supine) was calculated for each participant. Mean and standard deviation changes in heart rate (standing HR - supine HR) are reported for each study arm.
Measure: Mean (Standard Deviation); unit: beats/minute
Groups:
- POTS: Participants previously diagnosed with postural orthostatic tachycardia syndrome who were able to stand unassisted.
- Control-: Healthy volunteers that were free of chronic illness.
Arm/Group | POTS | Control-
Number analyzed (Participants) | 87 | 39
beats/minute | 15 (10) | 12 (8)

ADVERSE EVENTS:
Time Frame: During Study Visit, up to 1 hour
Description: Participants were not followed after study visit for adverse events.
Groups:
- POTS- Supine: Participants previously diagnosed with postural tachycardia syndrome age 13-60 years. Participants completed supine testing first, then standing.
- Control- Supine: Healthy volunteers with no chronic/systemic illness age 13-60 years. Participants completed supine testing first, then standing.
- POTS- Standing: Participants previously diagnosed with postural tachycardia syndrome age 13-60 years. Participants completed standing testing first, then supine.
- Control- Standing: Healthy volunteers with no chronic/systemic illness age 13-60 years.Participants completed standing testing first, then supine.
Arm/Group | POTS- Supine | Control- Supine | POTS- Standing | Control- Standing
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/139 | 0/139 | 0/139
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/139 | 0/139 | 0/139 | 0/139

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT03602482/Prot_SAP_000.pdf